CLINICAL TRIAL: NCT03562052
Title: LUng Cancer Screening With Low-dose Computed Tomography in a Population Exposed to Occupational Lung Carcinogens
Brief Title: Lung Cancer Screening in a Population Exposed to Occupational Lung Carcinogens
Acronym: LUCSO
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: University Hospital, Bordeaux (Other); Rennes University Hospital (Other); Centre Hospitalier Régional et Universitaire de Brest (Other); University Hospital, Caen (Other); University Hospital, Rouen (Other); Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: LUCSO
Record Dates: First submitted 2018-04-16; First posted 2018-06-19 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Lung Cancer
Keywords: Cancer; Lung; Occupational carcinogens; Tobacco smoking; Screening; Chest CT Scan; Asbestos
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Tobacco Smoking

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The good clinical practice guidelines for the surveillance of workers after occupational exposure to lung carcinogens were approved by the Haute Autorité de la Santé (French National Authority for Health) and the Institut National du Cancer (French National Cancer Institute) in December 2015 and one recommendation of these guidelines concerns the setting-up of a trial of low-dose chest computed tomography (CT) lung cancer screening in subjects occupationally exposed to lung carcinogens at high-risk of lung cancer (Expert consensus).

In LUCSO study, the investigators propose to conduct, under strictly defined conditions, a feasibility study of lung cancer screening in a population defined as being at high risk of lung cancer according to these good clinical practice guidelines. This population consists of smokers, aged from 55 to 74 years, currently or previously exposed to International Agency for Research on Cancer lung group 1 lung carcinogens.

The primary objective of this study is to evaluate the complex organization of lung cancer screening in the target population. This evaluation will focus on the following indicators:

* Screening activity indicator: screening coverage rate over two years
* Test quality indicator: validity of self-administered questionnaires to target the high-risk population
* Examination quality indicator: lung cancer detection rate, lung cancer detection rates by stage, validity of low-dose chest CT scan
* Follow-up indicator: smoking cessation rate, mortality rate This trial will be conducted in 8 French departments, by six reference centers specialized in occupational health (SRC).

In view of the exploratory nature of this trial, it is proposed to initially test the feasibility and acceptability of lung cancer screening sequentially over the first two years (Phase 1: 2021-2023, 24 months) in only two SRC (Val-de-Marne and Gironde).

The trial will be conducted in several steps:

1. Identification of subjects currently or previously occupationally exposed to lung carcinogens by a screening invitation letter sent by Departmental Cancer Screening Centers to subjects aged from 55 to 74 years.
2. Evaluation of occupational exposure to lung carcinogens
3. Evaluation of the lung cancer risk level and verification of eligibility
4. Screening procedure: Chest CT scans will be performed by centers specialized in chest imaging
5. Lung cancer follow-up when an abnormality suggestive of lung cancer is demonstrated.

DETAILED DESCRIPTION:
The good clinical practice guidelines for the surveillance of workers after occupational exposure to lung carcinogens were approved by the Haute Autorité de la Santé (French National Authority for Health) and the Institut National du Cancer (French National Cancer Institute) in December 2015 and the Recommendation R12 of these guidelines concerns the setting-up of a trial of low-dose chest computed tomography (CT) lung cancer screening in subjects occupationally exposed to lung carcinogens at high-risk of lung cancer (Expert consensus).

In LUCSO study, the investigators propose to conduct, under strictly defined conditions, a feasibility study of lung cancer screening in a population defined as being at high risk of lung cancer according to these good clinical practice guidelines. This population consists of smokers, aged from 55 to 74 years, currently or previously exposed to International Agency for Research on Cancer lung group 1 lung carcinogens.

The primary objective of this study is to evaluate the organization of lung cancer screening in the target population. This evaluation will focus on the following indicators:

* Screening activity indicator: screening coverage rate over two years
* Test quality indicator: validity of self-administered questionnaires to target the high-risk population
* Examination quality indicator: lung cancer detection rate, lung cancer detection rates by stage, validity of low-dose chest CT scan
* Follow-up indicator: smoking cessation rate, mortality rate

The secondary objectives of the study are:

* Describe the population recruited in each step of the protocol
* Develop a tool to identify subjects exposed to pulmonary carcinogens and with high-risk of lung cancer
* Evaluate the impact of the proposed screening programme on smoking cessation at one, two and three years.
* Evaluate the social impact of the screening campaign
* Conduct a cost-effectiveness analysis of the programme

The proposed study will take place in multidisciplinary and specialized reference centers (SRC) in various French districts participating in the programme, to welcome patients participating. It is organized into six workpackages (WP):

* WP1: Methodology - Epidemiology
* WP2: Evaluation of occupational exposure
* WP3: Imaging
* WP4: Lung cancer follow-up strategy
* WP5: Smoking cessation
* WP6: Medico-economic analysis Six specialized reference centers are proposed in four different regions in order to test a potential region effect and to allow the recruitment by each SRC of about 200 to 600 new eligible subjects per year and per department according to the population and the age pyramid of each department
* SRC1: Centre Intercommunal de Créteil for the Val-de-Marne (94), Seine-et-Marne (77), and Essonne (91) departments
* SRC2: Bordeaux University Hospital for the Gironde (33) department
* SRC3: Rennes University Hospital for the Ille-et-Vilaine (35) department
* SRC4: Brest University Hospital for the Finistère (29) department
* SRC5: Caen University Hospital for the Calvados (14) department
* SRC6: Rouen University Hospital for the Seine-Maritime (76) department

Each of these centers is voluntary and possesses the four essential prerequisites: an occupational health clinic - radiology team with specific skills in chest imaging - pulmonology team or network of pulmonologists specialized in lung cancer - smoking cessation team.

In view of the complexity of this organization, it is proposed to initially test the feasibility and acceptability of the screening programme sequentially for the first two years (24 months) in two SRCs (SRC1 and SRC2): "Phase 1: 2021-2023". It is expected to extend the study to the other SRCs after two years: "Phase 2: 2023-2029". Ad hoc adjustments will be decided for the creation of SRCs in the third year on the basis of the data acquired in the two pilot departments, especially on the expected target population participation rate. Mortality will be monitored at least until 2031.

The trial will be conducted in several steps:

1. Identification of subjects currently or previously occupationally exposed to lung carcinogens by a screening invitation letter sent by Departmental Cancer Screening Centers to subjects aged from 55 to 74 years.
2. Evaluation of occupational exposure to lung carcinogens
3. Evaluation of the lung cancer risk level and verification of eligibility
4. Screening procedure: Chest CT scans will be performed by centers specialized in chest imaging
5. Lung cancer follow-up when an abnormality suggestive of lung cancer is demonstrated.

ELIGIBILITY:
Inclusion Criteria:

Subjects at high risk of lung cancer: current smokers smoking 30 pack-years or more or ex-smokers smoking 30 pack-years or more and who have quit smoking for less than 15 years and currently or previously occupationally exposed to lung carcinogens. With an algorithm for determination of minimal duration of exposure to occupational carcinogens (according to the type and duration of occupational lung carcinogens)

Exclusion Criteria:

* Presence of clinical signs of lung cancer
* Subjects with a history of lung cancer
* Presence of serious short-term life-threatening comorbidities
* Absence of occupational exposure to lung carcinogens according to the predefined criteria
* Subjects already included in another prospective cohort study
* Subjects already assessed by chest CT scan during the previous year
* No tobacco exposure or insufficient tobacco exposure or smoking cessation for more than 15 years.

Ages: 55 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects aged from 55 to 74 years, current smokers smoking 30 pack-years or more or ex-smokers smoking 30 pack-years or more and who have quit smoking for less than 15 years and currently or previously occupationally exposed to lung carcinogens. These subjects are known to be high-risk population for lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2021-07-22 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2031-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of detected lung cancer | Year 1
  The proportion of subjects with lung cancer detected among the subjects performing the low-dose chest CT scan

SECONDARY OUTCOMES:
Rate of detected lung cancer | Year 2
  The proportion of subjects with lung cancer detected among the subjects performing the low-dose chest CT scan
Rate of detected lung cancer | Day 0
  The proportion of subjects with lung cancer detected among the subjects performing the low-dose chest CT scan
Participation rate | Day 0
  The proportion of subjects performing the low-dose chest CT scan among eligible responders during the first phase of the study
Rate of detected lung cancer in subjects exposed to occupational carcinogens | Day 0
  The proportion of subjects with lung cancer detected among the subjects exposed to occupational carcinogens and performing the low-dose chest CT scan
Rate of detected lung cancer in subjects exposed to occupational carcinogens | Year 1
  The proportion of subjects with lung cancer detected among the subjects exposed to occupational carcinogens and performing the low-dose chest CT scan
Rate of detected lung cancer in subjects exposed to occupational carcinogens | Year 2
  The proportion of subjects with lung cancer detected among the subjects exposed to occupational carcinogens and performing the low-dose chest CT scan
Stage of detected lung cancers | Day 0
Stage of detected lung cancers | Year 1
Stage of detected lung cancers | Year 2
Smoking cessation rate obtained in smokers in the sreened population | Year 3
  The proportion of subjects with smoking cessation among smokers
Mortality rate in the sreened population | Year 3
Mortality rate in the sreened population | Year 5
Mortality rate in the sreened population | Year 7
Mortality rate in the non-screened population | Year 3
Mortality rate in the non-screened population | Year 5
Lung cancer rate in non-screened subjects but met at the Occupational Disease Consultation Center | Year 3
Mortality rate in the non-screened population | Year 7
Lung cancer rate in non-screened subjects but met at the Occupational Disease Consultation Center | Year 5
Lung cancer rate in non-screened subjects but met at the Occupational Disease Consultation Center | Year 7
Rate of detected lung cancer and stage of detected lung cancer in the non-screened population | Year 3
Rate of detected lung cancer and stage of detected lung cancer in the non-screened population | Year 5
Rate of detected lung cancer and stage of detected lung cancer in the non-screened population | Year 7
Percentage of subjects participating in all screening (over the three years) | Year 3
Percentage of subjects participating in all screening (over the three years) | Year 4
Percentage of the subjects lost during follow-up in the screened population (follow-up at one year, two years, completion of other complementary exams) | Year 1
Percentage of the subjects lost during follow-up in the screened population (follow-up at one year, two years, completion of other complementary exams) | Year 2
Validity of the detailed personalised self-administered questionnaire for the evaluation of occupational exposures | Day 0
Number of cases recognized as occupational disease (for lung cancer or other occupational diseases) | Year 2
Proportion of invasive diagnostic procedures | Day 0
Proportion of invasive diagnostic procedures | Year 1
Proportion of invasive diagnostic procedures | Year 2
Proportion of non-invasive diagnostic procedures | Day 0
Proportion of non-invasive diagnostic procedures | Year 1
Proportion of non-invasive diagnostic procedures | Year 2
Proportion of serious and non-serious adverse events related to screening | Day 0
Proportion of serious and non-serious adverse events related to screening | Year 1
Proportion of serious and non-serious adverse events related to screening | Year 2
Proportion of subjects stopping smoking at each stage of screening | Day 0
Proportion of subjects stopping smoking at each stage of screening | Year 1
Proportion of subjects stopping smoking at each stage of screening | Year 2
The time period between each step of the screening (evaluation of the exposure, addressing in consultation of occupational diseases, inclusion, different exams of the follow-up) | Day 0
The time period between each step of the screening (evaluation of the exposure, addressing in consultation of occupational diseases, inclusion, different exams of the follow-up) | Year 1
The time period between each step of the screening (evaluation of the exposure, addressing in consultation of occupational diseases, inclusion, different exams of the follow-up) | Year 3
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Subject inclusion
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Year 1
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Year 2
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Year 3
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Year 4
Number of additional radiological examinations performed besides the prescribed CT scans of the protocol | Year 5
Number of hospitalizations | Subject inclusion
Number of hospitalizations | Year 1
Number of hospitalizations | Year 2
Number of hospitalizations | Year 3
Number of hospitalizations | Year 4
Number of hospitalizations | Year 5
Number of lung surgery | Subject inclusion
Number of lung surgery | Year 1
Number of lung surgery | Year 2
Number of lung surgery | Year 3
Number of lung surgery | Year 4
Number of lung surgery | Year 5
Number of chemotherapy | Day 0
Number of chemotherapy | Year 1
Number of chemotherapy | Year 2
Number of chemotherapy | Year 3
Number of chemotherapy | Year 4
Number of chemotherapy | Year 5

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Pairon, Pr, Principal Investigator — Centre Hospitalier Interconnmunal de Créteil
Locations (8):
- France (8):
  - Centre Hospitalier Universitaire de Bordeaux, Bordeaux
  - Université de Bordeaux, Bordeaux
  - Centre Hospitalier Universitaire de Brest, Brest
  - Centre Hospitalier Universitaire de Caen, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Universitaire de Rennes, Rennes
  - Centre Hospitalier Universitaire de Rouen, Rouen
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon

REFERENCES:
- [Derived] Delva F, Laurent F, Paris C, Belacel M, Brochard P, Bylicki O, Chouaid C, Clin B, Dewitte JD, Le Denmat V, Gehanno JF, Lacourt A, Margery J, Verdun-Esquer C, Mathoulin-Pelissier S, Pairon JC. LUCSO-1-French pilot study of LUng Cancer Screening with low-dose computed tomography in a smokers population exposed to Occupational lung carcinogens: study protocol. BMJ Open. 2019 Mar 23;9(3):e025026. doi: 10.1136/bmjopen-2018-025026. PMID 30904859